CLINICAL TRIAL: NCT06925906
Title: Characterizing Postoperative T and B Cell Dysfunction in Cancer Surgery Patients, Using COVID-19 as a Model Antigen
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: OHSNREB# 2011884-01H-CD8+-2025
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Abdominal Cancer
Keywords: Suppression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients with Abdominal cancers: Cancer patients who have been vaccinated with 2 or more doses of the Pfizer BNT162b1 vaccine

SUMMARY:
The Auer Lab research program studies how surgery affects the immune system and how this can lead to suppression in cancer patients which can lead to cancer reoccurrence. This has been well characterized in literature, with a clear demonstration that both surgery induced suppression of T cell and Natural Killer (NK) cell result in cancer recurrence..

The present study is the first in humans, to our knowledge, to demonstrate antigen specific dysfunction in T cells and B cells following cancer surgery. The study capitalized on the widespread vaccination of cancer patients against COVID before surgery, which allowed us to measure the response to the antigen S protein of SARS-CoV2. While the study is translational in methodology, we believe it will be of significant interest to all surgeons because it clearly establishes that surgery profoundly suppresses antigen-specific T and B cell responses, which have implications for postoperative infectious complications and cancer recurrence for those patients undergoing tumor resection

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of a primary abdominal malignancy consented to undergo major surgery with a planned length of stay of 3 or more days.
* Eligible patients must have signed a consent for surgical resection of the malignancy.
* Adequate hematological function defined as: platelet count ≥ 100 x 109/L, absolute neutrophil count ≥ 1 x 109/L, white blood count ≥ 2.5 x 109/L, hemoglobin count ≥ 90 g/L.
* Adequate organ functioning, including: total bilirubin ≤ 1.5 x upper limit of normal (ULN); AST, ALT < 2.5 x ULN; INR <1.5 ; CrCl>30mL/min.
* Ability to understand and provide a signed informed consent form (ICF) approved by the Institutional Review Board (IRB/IEC/REB).
* Ability to comply with protocol requirements.

Exclusion Criteria:

* Documented significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids, azathioprine, cyclosporin A). Subjects may be on physiologic doses of replacement prednisone or equivalent doses of corticosteroid (<7.5 mg daily).

  * History of autoimmune disease (even if controlled with medication) such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis.
  * Allergies or any contraindication to the use of tadalafil or any components of Cialis® or the influenza vaccine (including eggs), Agriflu®.
  * Serious intercurrent chronic or acute illness, or other illness considered by the investigator as an unwarranted high risk for an investigational product.
  * Patients who have suffered a myocardial infarction, stroke, or life-threatening arrhythmia within the last 6 months.
  * Patients with resting hypotension (BP <90/50 at rest) or hypertension (BP >170/110 at rest).
  * Patients with cardiac failure or coronary artery disease causing unstable angina.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ottawa Hospital Cancer patients undergoing abdominal surgeries
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-08-18 (Actual)

PRIMARY OUTCOMES:
Quantify the degree and determine the postoperative time course of antigen-specific T cell dysfunction following surgery | measured at day 0,1, 3, 28 post surgery
  Used the production of IFNγ, as measured by ELISpot, to determine the degree and duration of surgery-induced suppression of T cell responses to the RBD antigen.
Characterize the phenotype of dysfunctional CD8+ T cells in the immediate postoperative period | measured at day 0,1 post surgery
  Using multicolor flow cytometry, we characterized the cell surface markers, intracellular pathways and cytokines that are altered on POD1 in CD8+ T cells in response to RBD antigen.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Auer, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pre published article of the study. — https://www.biorxiv.org/content/10.1101/2024.12.23.629453v1